CLINICAL TRIAL: NCT05033080
Title: A Phase 3, Randomized, Double-blind, Controlled Study Evaluating the Efficacy and Safety of VX-121 Combination Therapy in Subjects With Cystic Fibrosis (CF) Who Are Heterozygous for F508del and a Minimal Function Mutation (F/MF)
Brief Title: A Phase 3 Study of VX-121 Combination Therapy in Participants With Cystic Fibrosis (CF) Heterozygous for F508del and a Minimal Function Mutation (F/MF)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX20-121-102; 2021-000712-31 (EudraCT Number)
Record Dates: First submitted 2021-08-26; First posted 2021-09-02 (Actual); Results first posted 2024-06-10 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-09

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — elexacaftor, ivacaftor, tezacaftor drug combination; ivacaftor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ELX/TEZ/IVA (Active Comparator): Following elexacftor/tezacaftor/ivacaftor (ELX/TEZ/IVA) run-in period of 4 weeks, participants received ELX 200 milligram (mg) once daily (qd) /TEZ 100 mg qd/IVA 150 mg every 12 hours (q12h) in the treatment period for 52 weeks.
  Interventions: Drug: ELX/TEZ/IVA; Drug: IVA; Drug: Placebo (matched to VX-121/TEZ/D-IVA)
- VX-121/TEZ/D-IVA (Experimental): Following ELX/TEZ/IVA run-in period of 4 weeks, participants received VX-121 20 mg qd/TEZ 100 mg qd/D-IVA 250 mg qd in the treatment period for 52 weeks.
  Interventions: Drug: VX-121/TEZ/D-IVA; Drug: Placebo (matched to ELX/TEZ/IVA); Drug: Placebo (matched to IVA)

INTERVENTIONS:
Drug: VX-121/TEZ/D-IVA — Fixed-dose combination tablets for oral administration.
  Other Names: VX-121/VX-661/CTP-656; VX-121/VX-661/VX-561; VX-121/tezacaftor/deutivacaftor
  Arms: VX-121/TEZ/D-IVA
Drug: ELX/TEZ/IVA — Fixed-dose combination tablets for oral administration.
  Other Names: VX-445/VX-661/VX-770; elexacaftor/tezacaftor/ivacaftor
  Arms: ELX/TEZ/IVA
Drug: IVA — Tablet for oral administration.
  Other Names: VX-770; ivacaftor
  Arms: ELX/TEZ/IVA
Drug: Placebo (matched to VX-121/TEZ/D-IVA) — Placebo matched to VX-121/TEZ/D-IVA for oral administration.
  Arms: ELX/TEZ/IVA
Drug: Placebo (matched to ELX/TEZ/IVA) — Placebo matched to ELX/TEZ/IVA for oral administration.
  Arms: VX-121/TEZ/D-IVA
Drug: Placebo (matched to IVA) — Placebo matched to IVA for oral administration.
  Arms: VX-121/TEZ/D-IVA

SUMMARY:
The purpose of this study evaluates the efficacy and safety of VX-121/tezacaftor/deutivacaftor (VX-121/TEZ/D-IVA) in CF participants who were heterozygous for F508del and a minimal function mutation (F/MF participants).

ELIGIBILITY:
Key Inclusion Criteria:

* Heterozygous for F508del and a minimal function mutation (F/MF genotype)
* Forced expiratory volume in 1 second (FEV1) value >=40% and <=90% of predicted mean for age, sex, and height for participants currently receiving ELX/TEZ/IVA therapy; FEV1 >=40% and <=80% for participants not currently receiving ELX/TEZ/IVA

Key Exclusion Criteria:

* History of solid organ or hematological transplantation
* Hepatic cirrhosis with portal hypertension, moderate hepatic impairment (Child Pugh Score 7 to 9), or severe hepatic impairment (Child Pugh Score 10 to 15)
* Lung infection with organisms associated with a more rapid decline in pulmonary status
* Pregnant or breast-feeding females

Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 435 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2023-05-12 (Actual); Study Completion 2023-11-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (139):
- United States (69):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Banner University of Arizona Medical Center, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Miller Children's Hospital / Long Beach Memorial, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Kaiser Permanente, Oakland, California
  - University of California Davis Medical Center, Sacramento, California
  - University of California San Francisco, Lung Transplant Program, San Francisco, California
  - Children's Hospital of Colorado, Aurora, Colorado
  - National Jewish Health, Denver, Colorado
  - University of Florida, Shands Hospital, Gainesville, Florida
  - Joe DiMaggio Cystic Fibrosis & Pulmonary Center, Hollywood, Florida
  - Central Florida Pulmonary Group, PA, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Johns Hopkins All Children's Hospital Outpatient Care Center, St. Petersburg, Florida
  - The Emory Clinic at Chantilly, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - St. Luke's Cystic Fibrosis Center of Idaho, Boise, Idaho
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Riley Hospital for Children at Indiana University Health, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Kosair Charities Pediatric Clinical Research Unit, Louisville, Kentucky
  - Tulane Medical Center, New Orleans, Louisiana
  - Massachusetts General Hospital Cystic Fibrosis Center Clinical Rsearch Center, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Michigan Medicine, Ann Arbor, Michigan
  - Helen DeVos Children's Hospital CF Center, Grand Rapids, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Childrens Hospital University of Missouri Health Sciences Center, Columbia, Missouri
  - The Children's Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Hospital - St. Louis University, St Louis, Missouri
  - Washington University School of Medicine / St. Louis Children's Hospital, St Louis, Missouri
  - Billings Clinic, Billings, Montana
  - Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth Hitchcock, Manchester, Manchester, New Hampshire
  - Morristown Medical Center, Morristown, New Jersey
  - Albany Medical College, Albany, New York
  - CF Therapeutics Development Center of Western New York, Buffalo, New York
  - Northwell Health- Long Island Jewish Medical Center, New Hyde Park, New York
  - Columbia University Medical Center, New York, New York
  - New York Medical College, Valhalla, New York
  - Atrium Health Levine Children's Hospital, Charlotte, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Cleveland Clinic CF, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Toledo Children's Hospital/Pediatric Pulmonary & Cystic Fibrosis Center, Toledo, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Sanford Children's Speciality Clinic, Sioux Falls, South Dakota
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Children's Foundation Research Center / Le Bonheur Children's Hospital, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - Cook Children's Health Care System, Fort Worth, Texas
  - Texas Children's Hospital - Baylor College of Medicine, Houston, Texas
  - University of Utah - Primary Children's Medical Center, Salt Lake City, Utah
  - Vermont Lung Center, Colchester, Vermont
  - University of Virginia Health System, Charlottesville, Virginia
  - Inova Fairfax, Falls Church, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- Australia (6):
  - Royal Prince Alfred Hospital, Camperdown
  - The Prince Charles Hospital, Chermside
  - Alfred Hospital, Melbourne, VIC
  - Mater Adult Hospital, South Brisbane
  - Queensland Children's Hospital, South Brisbane
  - Westmead Hospital, Westmead
- Czechia (2):
  - Klinika Detskych Infekcnich Nemoci, Brno
  - Fakultni nemocnice v Motole, Prague
- Germany (15):
  - Charite Paediatric Pulmonology Department, Berlin
  - St. Josef-Hospital, Bochum
  - Friedrich-Alexander University of Erlangen-Nuremberg, University Children's Hospital, Erlangen
  - Ruhrlandklinik Westdeutsches Lungenzentrum am Klinikum Essen, Essen
  - Universitatsklinikum Essen (AoR), Kinderklinik III, Abt. fur Pneumologie, Essen
  - Johann Wolfgang Goethe University, Frankfurt
  - Hannover Medical School, Hanover
  - Medizinische Hochschule Hannover, Hanover
  - Mukoviszidose-Zentrum am Universitätsklinikum Jena, Klinik für Kinder- und Jugendmedizin, Jena
  - Johannes Gutenberg-Universitaet, Mainz
  - Klinikum Innenstadt, University of Munich, München
  - Pneumologisches Studienzentrum Muenchen-West, München
  - Klinikum Westbrandenburg (CF), Potsdam
  - Universitätsklinikum Ulm, Klinik für Kinder- und Jugendmedizin (CF), Ulm
  - Universitätsklinikum Würzburg, Würzburg
- Hungary (2):
  - National Koranyi Institute for TBC and Pulmonology, Budapest
  - Pulmonology Institute Torokbalint, Törökbálint
- Ireland (7):
  - Cork University Hospital, Cork
  - Children's Health Ireland at Crumlin, Dublin
  - Children's Health Ireland at Tallaght, Dublin
  - Children's Health Ireland at Temple Street, Dublin
  - St. Vincent's University Hospital, Dublin
  - University Hospital Limerick (Adults), Limerick
  - University Hospital Limerick (Pediatrics), Limerick
- Israel (3):
  - Hadassah University Hospital Mount Scopus, Jerusalem
  - Schneider Children's Medical Center of Israel, Petach Tikvah
  - Sheba Medical Center - The Edmond and Lili Safra Children's Hospital, Tel Litwinsky
- New Zealand (4):
  - Greenlane Clinical Centre, Auckland
  - Starship Children's Hospital, Auckland
  - Canterbury Respiratory Research Group, Christchurch Hospital
  - Waikato Hospital, Hamilton
- Portugal (3):
  - Hospital de Santa Maria, Lisbon
  - CHP - Hospital de Santo Antonio, Porto
  - Hospital Sao Joao, Porto
- Spain (9):
  - Hospital Saint Joan de Deu, Barcelona
  - Hospital Universitari Vall d Hebron, Barcelona
  - Hospital Infantil Universitario Nino Jesus, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Virgen de la Arrixaca, Murcia
  - Corporacio Sanitaria Parc Tauli - Sabadell Hospital Universitari, Sabadell
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario y Politecnico La Fe, Valencia
- Sweden (3):
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Lund University Skanes Universitetssjukhus, Malmo
  - Karolinska Universitetssjukhuset, Huddinge, Stockholm
- United Kingdom (16):
  - Birmingham Heartlands Hospital, Birmingham
  - University Hospitals Bristol and Weston NHS Foundation Trust, Bristol Royal Hospital, Bristol
  - Royal Papworth Hospital NHS Foundation Trust, Cambridge
  - Royal Hospital for Sick Children, Edinburgh
  - Western General Hospital, Edinburgh
  - Royal Devon and Exeter Hospital, Exeter
  - Clinical Research Facility, Queen Elizabeth University Hospital, Glasgow
  - St. James University Hospital, Leeds
  - Liverpool Heart and Chest Hospital, Liverpool
  - King's College Hospital, London
  - Royal Brompton Hospital, London
  - St. Bartholomew's Hospital, London
  - Wythenshawe Hospital, Manchester
  - Clinical Research Facility, Newcastle upon Tyne
  - All Wales Adult Cystic Fibrosis Centre, University Hospital Llandough, Penarth
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing

REFERENCES:
- [Derived] Keating C, Yonker LM, Vermeulen F, Prais D, Linnemann RW, Trimble A, Kotsimbos T, Mermis J, Braun AT, O'Carroll M, Sutharsan S, Ramsey B, Mall MA, Taylor-Cousar JL, McKone EF, Tullis E, Floreth T, Michelson P, Sosnay PR, Nair N, Zahigian R, Martin H, Ahluwalia N, Lam A, Horsley A; VX20-121-102 Study Group; VX20-121-103 Study Group. Vanzacaftor-tezacaftor-deutivacaftor versus elexacaftor-tezacaftor-ivacaftor in individuals with cystic fibrosis aged 12 years and older (SKYLINE Trials VX20-121-102 and VX20-121-103): results from two randomised, active-controlled, phase 3 trials. Lancet Respir Med. 2025 Mar;13(3):256-271. doi: 10.1016/S2213-2600(24)00411-9. Epub 2025 Jan 2. PMID 39756424
- [Derived] Heneghan M, Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2023 Nov 20;11(11):CD010966. doi: 10.1002/14651858.CD010966.pub4. PMID 37983082

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in cystic fibrosis (CF) participants aged 12 years or older. It was pre-specified in the protocol to combine the data from this study with study VX20-121-103 (NCT05076149) for selected outcome measures.
Pre-assignment Details: A total of 435 participants were enrolled in this study, of which 37 were included in the run-in period but were not dosed in treatment period. Therefore, results are presented for only 398 participants dosed in the treatment period.
Period: Overall Study
Arm/Group | ELX/TEZ/IVA | VX-121/TEZ/D-IVA
Started | 202 | 196
Pooled Analysis Set (The Pooled full analysis set (PFAS) included all randomized participants from this study (VX20-121-102) and from Study VX20-121-103 who carry the intended CFTR genotype and received at least 1dose of study drug during the Treatment Period.) | 491 (Out of 491 participants, 202 participants were enrolled from this study and 289 participants were enrolled from VX20-121-103 study.) | 480 (Out of 480 participants,196 participants were enrolled from this study and 284 participants were enrolled from VX20-121-103 study.)
Completed | 191 | 184
Not Completed | 11 | 12
Not completed — Adverse Event | 4 | 4
Not completed — Withdrawal of consent (not due to AE) | 5 | 5
Not completed — Lost to Follow-up | 1 | 0
Not completed — Other non-compliance | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants who carry the intended CFTR genotype and received at least 1 dose of study drug in a study.
Groups:
- ELX/TEZ/IVA: Following ELX/TEZ/IVA run-in period of 4 weeks, participants received ELX 200 mg qd/TEZ 100 mg qd/IVA 150 mg q12h in the treatment period for 52 weeks.
- Total: Total of all reporting groups
Arm/Group | ELX/TEZ/IVA | VX-121/TEZ/D-IVA | Total
Number analyzed (Participants) | 202 | 196 | 398
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.9 (11.4) | 30.8 (10.5) | 30.8 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 80 | 163
  Male | 119 | 116 | 235
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 13 | 24
  Not Hispanic or Latino | 190 | 183 | 373
  Not Collected per Local Regulations | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 197 | 191 | 388
  Black or African American | 1 | 4 | 5
  Asian | 0 | 1 | 1
  Other | 1 | 0 | 1
  More than one race | 3 | 0 | 3
Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1) [Mean (Standard Deviation); unit: Percentage points] — FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration. Population: Here, "Number Analyzed" signifies participants who were evaluable for this study specific baseline measure. This analysis set (N=394) included participants who received the dose and who had a data for this efficacy analysis.
  Percentage points
    number analyzed (Participants) | 201 | 193 | 394
    (all) | 67.2 (14.6) | 67.0 (15.3) | 67.1 (15.0)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1)
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: From Baseline Through Week 24
Population: The Full Analysis Set (FAS) included all randomized participants who carried the intended CFTR mutation(s) and received at least 1 dose of study drug during Treatment Period. Here, "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage points
Arm/Group | ELX/TEZ/IVA | VX-121/TEZ/D-IVA
Number analyzed (Participants) | 193 | 187
percentage points | 0.3 [-0.3 to 0.9] | 0.5 [-0.1 to 1.1]
Statistical Analysis 1: Comparison: ELX/TEZ/IVA vs VX-121/TEZ/D-IVA; Test type: Non-Inferiority — The non-inferiority margin represents a clinically acceptable loss of effectiveness that margin preserve at least 50% of the treatment effect of the active control (ELX/TEZ/IVA) compared to placebo, where the treatment effect is estimated by the lower bound of the 95% confidence interval (CI); p < 0.0001, Mixed Models Repeated Measures; LS Mean difference = 0.2, 95% CI 2-sided [-0.7 to 1.1]

2. Secondary Outcome: Absolute Change in Sweat Chloride (SwCl)
Description: Sweat samples were collected using an approved collection device.
Time Frame: From Baseline Through Week 24
Population: FAS. Here, "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimole per liter (mmol/L)
Arm/Group | ELX/TEZ/IVA | VX-121/TEZ/D-IVA
Number analyzed (Participants) | 194 | 185
millimole per liter (mmol/L) | 0.9 [-0.6 to 2.3] | -7.5 [-9.0 to -6.0]
Statistical Analysis 1: Comparison: ELX/TEZ/IVA vs VX-121/TEZ/D-IVA; Test type: Superiority; p < 0.0001, Mixed Models Repeated Measures; LS Mean difference = -8.4, 95% CI 2-sided [-10.5 to -6.3]

3. Secondary Outcome: Percentage of Participants With SwCl <60 mmol/L (Pooled With Data From Study VX20-121-103)
Description: Sweat samples were collected using an approved collection device.
Time Frame: From Baseline Through Week 24
Population: The Pooled Full Analysis Set (PFAS) included all randomized participants from this study (VX20-121-102) and from Study VX20-121-103 who carried the intended CFTR mutation(s) and received at least 1 dose of study drug during the Treatment Period. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluated for this specific outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | ELX/TEZ/IVA | VX-121/TEZ/D-IVA
Number analyzed (Participants) | 479 | 465
percentage of participants | 76.6 | 85.8
Statistical Analysis 1: Comparison: ELX/TEZ/IVA vs VX-121/TEZ/D-IVA; Test type: Other; p < 0.0001, Generalized Estimated Equation Model; Odds Ratio (OR) = 2.21, 95% CI 2-sided [1.55 to 3.15]

4. Secondary Outcome: Percentage of Participants With SwCl <30 mmol/L (Pooled With Data From Study VX20-121-103)
Description: Sweat samples were collected using an approved collection device.
Time Frame: From Baseline Through Week 24
Population: PFAS. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluated for this specific outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | ELX/TEZ/IVA | VX-121/TEZ/D-IVA
Number analyzed (Participants) | 479 | 465
percentage of participants | 22.5 | 30.5
Statistical Analysis 1: Comparison: ELX/TEZ/IVA vs VX-121/TEZ/D-IVA; Test type: Other; p < 0.0001, Generalized Estimated Equation Model; Odds Ratio (OR) = 2.87, 95% CI 2-sided [2.00 to 4.12]

ADVERSE EVENTS:
Time Frame: Day 1 up to Safety follow-up (up to 56 weeks)
Description: Safety set include all participants who received at least 1 dose of study drug during the Treatment Period.
Groups:
- ELX/TEZ/IVA: Following ELX/TEZ/IVA run-in period of 4 weeks, participants received ELX 200 mg qd /TEZ 100 mg qd/IVA 150 mg q12h in the treatment period for 52 weeks.
- VNZ/TEZ/D-IVA: Following ELX/TEZ/IVA run-in period of 4 weeks, participants received VX-121 20 mg qd/TEZ 100 mg qd/D-IVA 250 mg qd in the treatment period for 52 weeks.
Arm/Group | ELX/TEZ/IVA | VNZ/TEZ/D-IVA
All-Cause Mortality (participants affected / at risk) | 0/202 | 0/196
Serious Adverse Events (participants affected / at risk) | 41/202 | 28/196
Other Adverse Events (participants affected / at risk) | 184/202 | 177/196
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ELX/TEZ/IVA (N=202) | VNZ/TEZ/D-IVA (N=196)
Arteriospasm coronary (Cardiac disorders) | 1 | 0
Cerebrovascular arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 0
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 1 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Mechanical ileus (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Subileus (Gastrointestinal disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 1
COVID-19 (Infections and infestations) | 3 | 1
Cellulitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 23 | 11
Influenza (Infections and infestations) | 1 | 3
Meningitis aseptic (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 1
Viral myocarditis (Infections and infestations) | 0 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Pulmonary function test decreased (Investigations) | 1 | 0
Hyperphosphatasaemia (Metabolism and nutrition disorders) | 0 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Serotonin syndrome (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 2
Behaviour disorder (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Depression suicidal (Psychiatric disorders) | 1 | 0
Mixed anxiety and depressive disorder (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ELX/TEZ/IVA (N=202) | VNZ/TEZ/D-IVA (N=196)
Abdominal distension (Gastrointestinal disorders) | 10 | 5
Abdominal pain (Gastrointestinal disorders) | 14 | 10
Abdominal pain upper (Gastrointestinal disorders) | 6 | 12
Diarrhoea (Gastrointestinal disorders) | 15 | 21
Nausea (Gastrointestinal disorders) | 17 | 7
Fatigue (General disorders) | 16 | 18
Pyrexia (General disorders) | 21 | 24
COVID-19 (Infections and infestations) | 53 | 49
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 64 | 53
Influenza (Infections and infestations) | 10 | 17
Nasopharyngitis (Infections and infestations) | 35 | 45
Respiratory tract infection (Infections and infestations) | 12 | 8
Sinusitis (Infections and infestations) | 10 | 10
Upper respiratory tract infection (Infections and infestations) | 27 | 17
Viral upper respiratory tract infection (Infections and infestations) | 18 | 17
Alanine aminotransferase increased (Investigations) | 10 | 13
Aspartate aminotransferase increased (Investigations) | 8 | 12
Blood creatine phosphokinase increased (Investigations) | 23 | 18
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 9
Headache (Nervous system disorders) | 22 | 25
Cough (Respiratory, thoracic and mediastinal disorders) | 41 | 45
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 10 | 13
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 24 | 19
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 23 | 24
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 | 12
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 14 | 19
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 14
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 21 | 18
Rash (Skin and subcutaneous tissue disorders) | 9 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-08-19): https://cdn.clinicaltrials.gov/large-docs/80/NCT05033080/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-18): https://cdn.clinicaltrials.gov/large-docs/80/NCT05033080/SAP_001.pdf